CLINICAL TRIAL: NCT06090266
Title: A Phase 1/2 Study of OR502 Alone and in Combination With Other Anti-cancer Agents in Subjects With Advanced Malignancies
Brief Title: A Study of OR502, a Monoclonal Antibody Targeting LILRB2, Alone and in Combination With Anticancer Agents
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoResponse, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR502-101
Record Dates: First submitted 2023-09-29; First posted 2023-10-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Tumor, Solid; Malignant Neoplasm; Metastatic Cancer; Advanced Solid Tumor; Cutaneous Melanoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OR502 monotherapy and combination therapy dose-escalation phase (Part A) (Experimental): Escalating repeated doses of OR502 by IV administration as monotherapy or in combination with cemiplimab in subjects with advanced solid tumors. OR502 will be administered once every 3 weeks (Q3W).
  Cemiplimab will be administered as an IV infusion at a dose of 350 mg.
  Interventions: Drug: OR502; Drug: Cemiplimab
- OR502 monotherapy and combination therapy dose-expansion phase (Part B) (Experimental): OR502 administered IV at 2 different dose levels identified in Part A as monotherapy or in combination with cemiplimab in subjects with platinum-resistant ovarian cancer and cutaneous squamous cell carcinoma.
  Cemiplimab will be administered as an IV infusion at a dose of 350 mg.
  Interventions: Drug: OR502; Drug: Cemiplimab

INTERVENTIONS:
Drug: OR502 — IgG1 monoclonal antibody that binds specifically to the LILRB2 protein.
Drug: Cemiplimab — IgG4 mAb that binds to PD-1 and blocks its interaction with PD-L1 and PD-L2.

SUMMARY:
This is an open-label, multicenter, first-in-human dose-escalation and expansion Phase 1-2 study designed to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of OR502 administered as a monotherapy and in combination with cemiplimab in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This Phase 1-2 study is designed to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of OR502, a fully human IgG1 antibody that binds specifically to LILRB2, in subjects with advanced solid tumors. The study consists parts:

Part A: a dose-escalation phase to determine the maximum-tolerated dose (MTD), maximum achievable dose, or optimal dose of OR502 for further evaluation as monotherapy and in combination with cemiplimab in a maximum of approximately 48 subjects. Recruitment closed.

Part B: an expansion phase in subjects with advanced solid tumors treated with OR502 at 2 separate doses as monotherapy followed by combination with cemiplimab, and in subjects with previously treated platinum-resistant ovarian cancer (PROC) or cutaneous squamous cell carcinoma (CSCC) treated with OR502 at 2 separate doses in combination with cemiplimab. Up to approximately 20 subjects will be treated in each arm of the 3 Part B cohorts to further characterize safety, help determine the recommended Phase 2 dose (RP2D) for further development and determine preliminary anti-tumor activity. Up to approximately 120 subjects total will be treated in Part B. Not yet open.

Part B4: a mini-expansion cohort in subjects with a histological diagnosis of cutaneous melanoma with advanced/metastatic disease. Subjects must have received a PD-(L)1 inhibitor-based therapy, either alone or in combination with other anti-cancer agents, for at least 12 weeks. Subjects in this cohort will be treated with OR502 as monotherapy. Actively recruiting.

Part B5: a mini-expansion cohort in subjects with a histological diagnosis of non-small cell lung cancer (NSCLC) with advanced/metastatic disease. Subjects must have received a PD-(L)1 inhibitor-based therapy, either alone or in combination with other anti-cancer agents, for at least 12 weeks. Subjects in this cohort will be treated with OR502 in combination with cemiplimab. Actively recruiting.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the subject prior to conducting study-specific procedures.
2. Male or female subjects ≥ 18 years of age.
3. Histological diagnosis as follows:

   1. Parts A and B (Cohorts A1, A2, and B1): subjects must have a histological diagnosis of any type of carcinoma, sarcoma, or melanoma with progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy with curative intent.
   2. Part B (Expansion Cohorts B2-B3): subjects must have a histological diagnosis of the relevant tumor type (CSCC or PROC) with advanced/metastatic disease not amenable to local therapy with curative intent.
4. Prior therapies:

   a. Part A (dose-escalation) and Cohort B1 (monotherapy expansion) i. Subjects must have experienced progressive disease (PD) on an established standard systemic anti-cancer therapy for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds. Subjects must have no available proven curative or life prolonging therapies.

   b. Cohorts B4 and B5 (mini-expansion cohorts) i. Subjects must have received a PD-(L)1 inhibitor-based therapy, either alone or in combination with other anti-cancer agents, for at least 12 weeks. If subjects have received other lines of immunotherapy, including PD-(L)1-based therapy, they must have demonstrated clinical benefit on each prior immunotherapy. Subjects may also have received additional anti-cancer therapies after failure of a PD-(L)1 inhibitor, but 2nd line subjects are preferred.

   c. Cohorts B2 and B3 (dose-expansion) i. Cohort B2 subjects (CSCC) must have received a PD-(L)1 inhibitor. Subjects may not have received an additional immunotherapy.

   ii. Cohort B3 subjects (PROC) must have received platinum-based therapy and experienced disease progression on or within 6 months of completion of such therapy. Subjects may have received prior anti-PD-1 therapy. Subjects may have received additional therapies after failure of platinum-based therapy.
5. Subjects must have measurable disease per RECIST v1.1.
6. People of childbearing potential, if not postmenopausal (defined as no menses for at least 12 continuous months prior to study entry) or surgically sterile, must be willing to practice at least one of the highly effective methods of birth control described in Section 4.3 for at least a menstrual cycle (or partner's menstrual cycle, for male subjects) before and for 4 months after study medication administration.
7. Resolution of prior clinically significant therapy-related AEs (excluding alopecia and ≤ Grade 2 peripheral neuropathy) to ≤ Grade 1 per NCI-CTCAE version 5.0, and no treatment for these AEs for at least 2 weeks prior to the time of enrollment. Electrolyte and hormonal supplementation may be used to treat these AEs provided the subject is stable on these supplements.
8. Minimum of 2 weeks since the last dose of other hormone therapy and 3 weeks since the last dose of other systemic cancer therapy or radiotherapy (> 4 weeks in case of nitrosoureas or radio-immuno conjugate therapy). Adjuvant hormonal therapy (e.g., tamoxifen) is allowed provided the original tumor diagnosis was more than 3 years before the first dose of study medication. Subjects with prostate cancer on stable doses of anti-hormone treatment may remain on therapy for this trial.
9. Subjects must have adequate organ function.
10. Biopsy specimens:

    1. All subjects must be able to supply an archival tumor tissue specimen. If an archival specimen is not available, subjects may remain eligible with approval of the medical monitor.
    2. Subjects in Cohort B1 must consent to pre- and on-treatment biopsies. Tissue obtained for the biopsy must not be previously irradiated. No systemic anti-neoplastic therapy may be received by the subject between the time of the biopsy and the first administration of study medication.
    3. Subjects in all other cohorts will be asked to consent to pre- and on-treatment biopsies for biomarker analysis of the acquired tissue. These biopsies are optional and not required for study participation. Tissue obtained for the biopsy must not be previously irradiated. No systemic anti-neoplastic therapy may be received by the subject between the time of the biopsy and the first administration of study medication.
11. Subject is able and willing to comply with the protocol and the restrictions and assessments therein.
12. As required by local regulations or law, subjects must fulfill the obligation of affiliation or beneficiary of a social security or similar scheme.

Exclusion Criteria:

1. Subject previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
2. Life expectancy < 12 weeks.
3. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) > 2.
4. Prior organ or stem cell transplant.
5. Subjects with symptomatic ascites or pleural effusion. Subjects who are clinically stable for at least 2 weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis) are eligible.
6. Subject has a known active central nervous system (CNS) primary tumor or metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no radiological evidence of new or enlarging brain metastases, and are off steroids or on a stable dose up to an equivalent of prednisone 10 mg/day for at least 15 days prior to first dose of study medication. Subjects who have symptoms consistent with CNS metastasis must have a negative magnetic resonance imaging (MRI) scan during the screening period.
7. Subject has a known history of a hematologic malignancy, malignant primary brain tumor, or another malignant primary solid tumor (other than that under study), unless the subject has undergone potentially curative therapy with no evidence of recurrent disease for at least 3 years before the start of treatment.

   1. Subjects with a known history of AJCC Stage 1 cancer that has undergone potentially curative therapy with no evidence of recurrent disease for at least 1 year before the start of treatment may be eligible at the Investigator's discretion after consultation with the Sponsor.
   2. Subjects who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers at any time before the start of treatment, and have no evidence of recurrent disease, are eligible.
8. Recent or ongoing serious infection including the following:

   1. Any uncontrolled Grade 3 or higher (per NCI-CTCAE version 5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of OR502. Routine antimicrobial prophylaxis is allowed.
   2. Uncontrolled infection with human immunodeficiency virus (HIV). Subjects on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
   3. Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for hepatitis B indicating acute or chronic infection. Subjects who are or have received anti-HBV therapy and have undetectable HBV DNA for at least 6 months prior to study entry are eligible. Serological testing for hepatitis B at screening is not required.
   4. Known active hepatitis C as determined by positive serology and confirmed by polymerase chain reaction (PCR). Subjects on or having received anti-retroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for hepatitis C at screening is not required.
   5. Known active or latent tuberculosis (testing at screening is not required).
9. Autoimmune disease or inflammatory condition requiring systemic anti-inflammatory therapy with exceptions as noted in Exclusion Criterion 10. Subjects on hormone replacement therapy for autoimmune-induced endocrinopathies are eligible.
10. Use of systemic corticosteroids within 15 days or other immunosuppressive drugs within 30 days prior to start of the study, with the exception of corticosteroids as replacement therapy up to an equivalent of prednisone 10 mg/day, which are allowed.
11. QTc interval ≥ 470 msec by electrocardiogram (ECG).
12. Subject has received an investigational product or been treated with an investigational device within 30 days prior to first administration of study medication.
13. Subject has received a live vaccine within 30 days prior to first administration of study medication.
14. For Cohorts A2, B1, B2, and B3 only:

    1. Known hypersensitivity to cemiplimab or any of its excipients or contraindicated to cemiplimab per approved local labeling.
    2. Interstitial lung disease.
    3. Prior pneumonitis requiring systemic corticosteroid therapy.
    4. Receiving immunosuppressive therapy, with exceptions as noted in Exclusion Criterion 10.
    5. A history of severe immune-related adverse reactions from treatment with ipilimumab, defined as any Grade 4 toxicity or Grade 3 toxicity requiring corticosteroid treatment (> 10 mg/day prednisone or equivalent) for more than 12 weeks.
15. Concurrent therapy with anti-cancer or anti-neoplastic drugs, with the exception of adjuvant hormonal therapy, which is allowed as outlined in Inclusion Criterion 8.
16. History or clinical evidence of any surgical or medical condition that the Investigator judges as likely to interfere with the results of the study or pose an additional risk in participating, e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, autoimmune or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
17. Subjects who, at the time of signing informed consent, had a recent history (within the last year) of chronic substance abuse.
18. Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
19. Vulnerable persons: subjects under judicial safeguard, subjects deprived of their liberty by judicial or administrative decision, subjects under psychiatric care without their consent, subjects admitted to a health or social institution for purposes other than research, adults subject to a measure of legal protection (guardianship or curatorship), and subjects unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Adverse Events and Serious Adverse Events | Screening to 90 days from last dose.
  The nature, frequency, and severity of adverse events and serious adverse events graded by CTCAE v 5.0 as aggregated descriptive findings.
Vital Signs | Screening to 90 days from last dose.
  Assessment of changes in vital sign measurements (heart rate, pulse oximetry and blood pressure) as aggregated descriptive findings.
Recommended Dose and Regimen (mono and combination therapy) | Screening to 90 days from last dose.
  Determination of the recommended dose of OR502 for further development.

SECONDARY OUTCOMES:
Pharmacokinetics of OR502 | Day 1 of dosing through 21 days post last dose.
  Peak plasma concentration (Cmax).
Pharmacokinetics of OR502 | Day 1 of dosing through 21 days post last dose.
  Area under the plasma concentration versus time curve (AUC).
Objective Response Rate (ORR) | Day 1 of dosing through 90 days after the last dose.
  ORR according to RECIST v1.1.
Disease Control Rate (DCR) | Day 1 of dosing through 90 days after the last dose.
  The percentage of subjects with a complete response, partial response, or stable disease for at least 2 consecutive tumor assessments.
Progression Free Survival (PFS) | Day 1 of dosing through 90 days after the last dose.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for PD or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NEXT Austin, Austin, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No